CLINICAL TRIAL: NCT03149822
Title: Phase I/II Study of Pembrolizumab and Cabozantinib in Patients With Metastatic Renal Cell Carcinoma
Brief Title: Study of Pembrolizumab and Cabozantinib in Patients With Metastatic Renal Cell Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 16-2300.cc; NCI-2017-01777 (Other: CTRP)
Record Dates: First submitted 2017-04-28; First posted 2017-05-11 (Actual); Results first posted 2023-10-17 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Metastatic Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — cabozantinib; pembrolizumab

STUDY DESIGN:
Masking Description: Open-Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Phase 1: Pembrolizumab 200 mg plus Cabozantinib 40mg (Experimental): Pembrolizumab 200 mg intravenous (IV) infusion on day 1 of each 21-day cycle in combination with cabozantinib 40 mg orally once daily until disease progression, unacceptable toxicity, or consent withdrawal.
  Interventions: Drug: Cabozantinib; Drug: Pembrolizumab
- Phase 1: Pembrolizumab 200 mg plus Cabozantinib 60mg (Experimental): Pembrolizumab 200 mg intravenous (IV) infusion on day 1 of each 21-day cycle in combination with cabozantinib 60 mg orally once daily until disease progression, unacceptable toxicity, or consent withdrawal.
  Interventions: Drug: Cabozantinib; Drug: Pembrolizumab
- Phase 2: Pembrolizumab 200 mg plus Cabozantinib at the RP2D (Experimental): Pembrolizumab 200 mg intravenous (IV) infusion on day 1 of each 21-day cycle in combination with cabozantinib at the RP2D orally once daily for up to 35 cycles, until disease progression, unacceptable toxicity, or consent withdrawal. All participants who stop pembrolizumab after 35 cycles with SD or better may be eligible for up to an additional 17 cycles (approximately 1 year) of pembrolizumab treatment if they progress after stopping pembrolizumab from the initial treatment phase.
  Interventions: Drug: Cabozantinib; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Cabozantinib — Pharmaceutical form: tablets Route of administration: oral
  Other Names: Cabometyx
Drug: Pembrolizumab — Pharmaceutical form: solution Route of administration: injection
  Other Names: MK-3475; Keytruda

SUMMARY:
This is a phase I/II open-label study designed to evaluate the combination of pembrolizumab and cabozantinib in subjects with locally advanced, recurrent, or metastatic renal cell carcinoma. Sequential dose escalation of cabozantinib with standard dose pembrolizumab will occur in the phase I dose escalation part of the study to determine the recommended phase 2 dose (RP2D). Subsequently, subjects will receive cabozantinib at the RP2D in combination with pembrolizumab in the phase II dose expansion part of the study.

DETAILED DESCRIPTION:
Primary Objectives

* To determine the efficacy based on objective response rate [ORR = complete response (CR) + partial response (PR)] of pembrolizumab and cabozantinib when administered in combination in subjects with locally advanced or metastatic renal cell carcinoma..

Secondary Objectives

* To characterize dose-limiting toxicities (DLTs), maximum tolerated dose (MTD), and recommended phase 2 dose (RP2D) for the combination.
* To assess other measures of anti-tumor activity of the combination of pembrolizumab and cabozantinib in subjects with locally advanced or metastatic renal cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have histological or cytological documentation of renal cell carcinoma
2. Subjects must have locally advanced, recurrent, or metastatic disease.
3. Be willing and able to provide written informed consent/assent for the trial.
4. Stated willingness to complywith all study procedures and be available for the duration of the trial.
5. Be ≥ 18 years of age on day of signing informed consent.
6. Have measurable or evaluable disease based on RECIST 1.1.
7. Recovery to baseline or ≤ Grade 1 CTCAE v.4.0 from toxicities related to any prior treatments, unless AE(s) are clinically non-significant and/or stable on supportive therapy.
8. Confirmed availability of representative archival tumor specimens in paraffin blocks (preferred) or ≥ 10 unstained slides, with an associated pathology report.

   * Acceptable samples include core needle biopsies for deep tumor tissue or excisional, incisional, or punch biopsies for cutaneous, subcutaneous, or mucosal lesions.
   * Tumor tissue from bone metastases is not evaluable for PD-L1 expression and is therefore not acceptable.
   * A subject with insufficient or unavailable archival tissue may be eligible, upon discussion with the Principal Investigator, if the subject is willing to consent to undergo a pretreatment core, punch, or excisional/incisional biopsy sample collection of the tumor.
9. Have a performance status of 0 or 1 on the ECOG Performance Scale.
10. Demonstrate adequate organ function as defined by desired lab values.
11. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
12. Female subjects of childbearing potential (Section 5.7.2) must be willing to use an adequate method of contraception as outlined in Section 5.7.2 - Contraception, for the course of the study through 120 days after the last dose of study medication. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
13. Male subjects of childbearing potential (Section 5.7.1) must agree to use an adequate method of contraception as outlined in Section 5.7.1- Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroiderapy equivalent to ≥ 10 mg/day of prednisone, or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Has a known history of active TB (Bacillus Tuberculosis)
4. Has had prior treatment with pembrolizumab.
5. Has had prior treatment with cabozantinib.
6. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.

   - Note: Subjects with stable, treated hypothyroidism or adrenal insufficiency may qualify for the study
7. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Subjects with hypertension managed with medication are an exception to this criterion and may qualify for the study.
   * Subjects with ≤ Grade 2 endocrinopathy (e.g. hypothyroidism or adrenal insufficiency managed with medication) are an exception to this criterion and may qualify for the study.
8. Has had major surgery within 4 weeks or minor surgery within 2 weeks prior to study Day 1. Subjects must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
9. Prior treatment with immune checkpoint inhibitors is allowed, provided that no treatment-related Grade ≥ 3 adverse events (other than Grade 3 endocrinopathy managed with replacement therapy) were observed and at least a minimum of 28 days have elapsed between the last dose of prior treatment and the proposed Cycle 1 Day 1.
10. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer, carcinoma in situ or superficial bladder cancer, low-grade prostate cancer, intraductal papillary mucinous neoplasm (IPMN), and other low grade cancers that is suitable for active surveillance in the opinion of the investigator.
11. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Active CNS metastases will be defined as brain lesions that 1) require intervention with surgery, stereotactic radiosurgery (SRS), or whole brain radiotherapy (WBRT) or 2) require anti-epileptic therapy, systemic steroid treatment, or intrathecal therapy. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks after completion of focal therapy for brain metastases and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis, which is excluded regardless of clinical stability.
12. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is allowed.
13. Has history of solid organ transplantation.
14. Has history of osteonecrosis of the jaw.
15. Has history of reversible posterior leukoencephalopathy syndrome.
16. Has history of wound dehiscence or complications requiring medical intervention within 6 months of study entry.
17. Has history of (non-infectious) pneumonitis that required steroids or active, non- infectious pneumonitis.
18. Has an active infection requiring systemic therapy with IV antibiotics.
19. Has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

    1. Cardiovascular disorders:

       * Symptomatic congestive heart failure, unstable angina pectoris, serious cardiac arrhythmias.
       * Uncontrolled hypertension defined as sustained BP > 150 mm Hg systolic or > 100 mm Hg diastolic despite optimal antihypertensive treatment.
       * Stroke (including TIA), myocardial infarction, or other ischemic event, or thromboembolic event (e.g., deep venous thrombosis, pulmonary embolism) within 3 months before randomization.
    2. Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation:

       * Tumors invading the GI-tract, active peptic ulcer disease, inflammatory bowel disease, diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis or acute obstruction of the pancreatic or biliary duct, or gastric outlet obstruction.
       * Abdominal fistula, gastrointestinal perforation, bowel obstruction, or intra-abdominal abscess within 6 months before randomization. Complete healing of an intra-abdominal abscess must be confirmed before study initiation.
    3. Has clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon within 3 months before randomization.
    4. Known endobronchial disease manifestation. Patients with suspected endobronchial disease on imaging who have no evidence of endobronchial disease on bronchoscopy are allowed. Patients with treated endobronchial disease are also allowed provided they are stable.
    5. Lesions invading major pulmonary blood vessels.
20. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
21. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
22. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
23. Has an inability to swallow tablets or capsules.
24. Has a previously identified allergy or hypersensitivity to components of the study treatment formulations.
25. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
26. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
27. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2024-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Lam, MD, Principal Investigator — University of Colorado, Denver
Locations (5):
- United States (5):
  - University of Colorado Denver, Aurora, Colorado
  - Memorial Hospital Central, Colorado Springs, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Highlands Ranch Hospital, Highlands Ranch, Colorado
  - UCHealth Lone Tree Medical Center, Lone Tree, Colorado

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gunturi A, McDermott DF. Potential of new therapies like anti-PD1 in kidney cancer. Curr Treat Options Oncol. 2014 Mar;15(1):137-46. doi: 10.1007/s11864-013-0268-y. PMID 24504486
- [Background] Philips GK, Atkins MB. New agents and new targets for renal cell carcinoma. Am Soc Clin Oncol Educ Book. 2014:e222-7. doi: 10.14694/EdBook_AM.2014.34.e222. PMID 24857106
- [Background] Hato T, Zhu AX, Duda DG. Rationally combining anti-VEGF therapy with checkpoint inhibitors in hepatocellular carcinoma. Immunotherapy. 2016;8(3):299-313. doi: 10.2217/imt.15.126. Epub 2016 Feb 11. PMID 26865127
- [Background] Massari F, Santoni M, Ciccarese C, Santini D, Alfieri S, Martignoni G, Brunelli M, Piva F, Berardi R, Montironi R, Porta C, Cascinu S, Tortora G. PD-1 blockade therapy in renal cell carcinoma: current studies and future promises. Cancer Treat Rev. 2015 Feb;41(2):114-21. doi: 10.1016/j.ctrv.2014.12.013. Epub 2015 Jan 6. PMID 25586601
- [Background] Motzer RJ, Escudier B, McDermott DF, George S, Hammers HJ, Srinivas S, Tykodi SS, Sosman JA, Procopio G, Plimack ER, Castellano D, Choueiri TK, Gurney H, Donskov F, Bono P, Wagstaff J, Gauler TC, Ueda T, Tomita Y, Schutz FA, Kollmannsberger C, Larkin J, Ravaud A, Simon JS, Xu LA, Waxman IM, Sharma P; CheckMate 025 Investigators. Nivolumab versus Everolimus in Advanced Renal-Cell Carcinoma. N Engl J Med. 2015 Nov 5;373(19):1803-13. doi: 10.1056/NEJMoa1510665. Epub 2015 Sep 25. PMID 26406148
- [Background] Ko JS, Zea AH, Rini BI, Ireland JL, Elson P, Cohen P, Golshayan A, Rayman PA, Wood L, Garcia J, Dreicer R, Bukowski R, Finke JH. Sunitinib mediates reversal of myeloid-derived suppressor cell accumulation in renal cell carcinoma patients. Clin Cancer Res. 2009 Mar 15;15(6):2148-57. doi: 10.1158/1078-0432.CCR-08-1332. Epub 2009 Mar 10. PMID 19276286
- [Background] Tartour E, Pere H, Maillere B, Terme M, Merillon N, Taieb J, Sandoval F, Quintin-Colonna F, Lacerda K, Karadimou A, Badoual C, Tedgui A, Fridman WH, Oudard S. Angiogenesis and immunity: a bidirectional link potentially relevant for the monitoring of antiangiogenic therapy and the development of novel therapeutic combination with immunotherapy. Cancer Metastasis Rev. 2011 Mar;30(1):83-95. doi: 10.1007/s10555-011-9281-4. PMID 21249423
- [Background] Terme M, Colussi O, Marcheteau E, Tanchot C, Tartour E, Taieb J. Modulation of immunity by antiangiogenic molecules in cancer. Clin Dev Immunol. 2012;2012:492920. doi: 10.1155/2012/492920. Epub 2012 Dec 24. PMID 23320019
- [Background] Voron T, Colussi O, Marcheteau E, Pernot S, Nizard M, Pointet AL, Latreche S, Bergaya S, Benhamouda N, Tanchot C, Stockmann C, Combe P, Berger A, Zinzindohoue F, Yagita H, Tartour E, Taieb J, Terme M. VEGF-A modulates expression of inhibitory checkpoints on CD8+ T cells in tumors. J Exp Med. 2015 Feb 9;212(2):139-48. doi: 10.1084/jem.20140559. Epub 2015 Jan 19. PMID 25601652
- [Background] Carmeliet P, Jain RK. Principles and mechanisms of vessel normalization for cancer and other angiogenic diseases. Nat Rev Drug Discov. 2011 Jun;10(6):417-27. doi: 10.1038/nrd3455. PMID 21629292
- [Background] Nickerson ML, Jaeger E, Shi Y, Durocher JA, Mahurkar S, Zaridze D, Matveev V, Janout V, Kollarova H, Bencko V, Navratilova M, Szeszenia-Dabrowska N, Mates D, Mukeria A, Holcatova I, Schmidt LS, Toro JR, Karami S, Hung R, Gerard GF, Linehan WM, Merino M, Zbar B, Boffetta P, Brennan P, Rothman N, Chow WH, Waldman FM, Moore LE. Improved identification of von Hippel-Lindau gene alterations in clear cell renal tumors. Clin Cancer Res. 2008 Aug 1;14(15):4726-34. doi: 10.1158/1078-0432.CCR-07-4921. PMID 18676741
- [Background] Gibney GT, Aziz SA, Camp RL, Conrad P, Schwartz BE, Chen CR, Kelly WK, Kluger HM. c-Met is a prognostic marker and potential therapeutic target in clear cell renal cell carcinoma. Ann Oncol. 2013 Feb;24(2):343-349. doi: 10.1093/annonc/mds463. Epub 2012 Sep 28. PMID 23022995
- [Background] Mukai S, Yorita K, Kawagoe Y, Katayama Y, Nakahara K, Kamibeppu T, Sugie S, Tukino H, Kamoto T, Kataoka H. Matriptase and MET are prominently expressed at the site of bone metastasis in renal cell carcinoma: immunohistochemical analysis. Hum Cell. 2015 Jan;28(1):44-50. doi: 10.1007/s13577-014-0101-3. Epub 2014 Sep 4. PMID 25186085
- [Background] Schiefer AI, Mesteri I, Berghoff AS, Haitel A, Schmidinger M, Preusser M, Birner P. Evaluation of tyrosine kinase receptors in brain metastases of clear cell renal cell carcinoma reveals cMet as a negative prognostic factor. Histopathology. 2015 Dec;67(6):799-805. doi: 10.1111/his.12709. Epub 2015 Jun 7. PMID 25847631
- [Background] Sutherland DE, Morrow CE, Florack G, Kretschmer GJ, Baumgartner D, Matas AJ, Najarian JS. Cold storage preservation of islet and pancreas grafts as assessed by in vivo function after transplantation to diabetic hosts. Cryobiology. 1983 Apr;20(2):138-50. doi: 10.1016/0011-2240(83)90003-2. No abstract available. PMID 6406150
- [Background] Choueiri TK, Halabi S, Sanford BL, Hahn O, Michaelson MD, Walsh MK, Feldman DR, Olencki T, Picus J, Small EJ, Dakhil S, George DJ, Morris MJ. Cabozantinib Versus Sunitinib As Initial Targeted Therapy for Patients With Metastatic Renal Cell Carcinoma of Poor or Intermediate Risk: The Alliance A031203 CABOSUN Trial. J Clin Oncol. 2017 Feb 20;35(6):591-597. doi: 10.1200/JCO.2016.70.7398. Epub 2016 Nov 14. PMID 28199818
- [Background] Harshman LC, Choueiri TK. Targeting the hepatocyte growth factor/c-Met signaling pathway in renal cell carcinoma. Cancer J. 2013 Jul-Aug;19(4):316-23. doi: 10.1097/PPO.0b013e31829e3c9a. PMID 23867513
- [Background] Choueiri TK, Pal SK, McDermott DF, Morrissey S, Ferguson KC, Holland J, Kaelin WG, Dutcher JP. A phase I study of cabozantinib (XL184) in patients with renal cell cancer. Ann Oncol. 2014 Aug;25(8):1603-8. doi: 10.1093/annonc/mdu184. Epub 2014 May 14. PMID 24827131
- [Derived] Kessler ER, Callihan E, Hu J, Eule C, Srivastava G, Kemme DJ, Iruku P, Rana V, Moore J, Schuster SR, Amirault M, Flaig TW, Lam ET. A Phase I/II Clinical Trial of Pembrolizumab and Cabozantinib in Metastatic Renal Cell Carcinoma. Cancer Res Commun. 2023 Jun 8;3(6):1004-1012. doi: 10.1158/2767-9764.CRC-23-0060. eCollection 2023 Jun. PMID 37377613

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Phase 1: Pembrolizumab 200 mg Plus Cabozantinib 40mg | Phase 1: Pembrolizumab 200 mg Plus Cabozantinib 60mg | Phase 2: Pembrolizumab 200 mg Plus Cabozantinib at the RP2D
Started | 5 | 3 | 37
Completed | 5 | 3 | 37
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1: Pembrolizumab 200 mg Plus Cabozantinib 40mg | Phase 1: Pembrolizumab 200 mg Plus Cabozantinib 60mg | Phase 2: Pembrolizumab 200 mg Plus Cabozantinib at the RP2D | Total
Number analyzed (Participants) | 5 | 3 | 37 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 20 | 27
  >=65 years | 1 | 0 | 17 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (9.8) | 48.7 (9.6) | 61.7 (11.5) | 60.1 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 10 | 12
  Male | 3 | 3 | 27 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 5 | 3 | 33 | 41
  Unknown or Not Reported | 0 | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 3 | 3
  White | 5 | 3 | 32 | 40
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 5 | 3 | 37 | 45

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Pembrolizumab and Cabozantinib Based on Objective Response Rate
Description: Measured through the complete response (CR) + partial response (PR)] of pembrolizumab and cabozantinib when administered in combination in subjects with locally advanced or metastatic renal cell carcinoma. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Beginning of study to end of study, up to 5 years
Population: Total RCC patients who were evaluable for response at the dose level
Measure: Number (95% Confidence Interval); unit: % of patients
Groups:
- Phase 1/2: All Evaluable Patients Treated at Pembrolizumab 200 mg IV Q3W + Cabozantinib 60 mg PO QD: Pembrolizumab 200 mg intravenous (IV) infusion on day 1 of each 21-day cycle in combination with cabozantinib at the RP2D orally once daily for up to 35 cycles, until disease progression, unacceptable toxicity, or consent withdrawal. All participants who stop pembrolizumab after 35 cycles with SD or better may be eligible for up to an additional 17 cycles (approximately 1 year) of pembrolizumab treatment if they progress after stopping pembrolizumab from the initial treatment phase.
  Cabozantinib: Pharmaceutical form: tablets Route of administration: oral
  Pembrolizumab: Pharmaceutical form: solution Route of administration: injection
- Phase 1 Dose Escalation Cohort: Pembrolizumab 200 mg IV Q3W Plus Cabozantinib 40mg PO QD: Pembrolizumab 200 mg intravenous (IV) infusion on day 1 of each 21-day cycle in combination with cabozantinib 40 mg orally once daily until disease progression, unacceptable toxicity, or consent withdrawal.
  Cabozantinib: Pharmaceutical form: tablets Route of administration: oral
  Pembrolizumab: Pharmaceutical form: solution Route of administration: injection
Arm/Group | Phase 1/2: All Evaluable Patients Treated at Pembrolizumab 200 mg IV Q3W + Cabozantinib 60 mg PO QD | Phase 1 Dose Escalation Cohort: Pembrolizumab 200 mg IV Q3W Plus Cabozantinib 40mg PO QD
Number analyzed (Participants) | 38 | 5
% of patients | 65.8 [49.9 to 78.8] | 0 [0 to 0]

2. Secondary Outcome: Maximally Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D)
Description: * The MTD is defined as the highest dose level with no more than 1 DLT reported in 6 DLT-evaluable subjects.
  * The Recommended Phase 2 Dose (RP2D) of cabozantinib will be selected based on the clinical data and will not exceed the MTD. If < 2/6 subjects experience a DLT at 60 mg daily during dose escalation, then 60 mg daily will be considered the RP2D. If ≥ 2/6 subjects experience DLTs at 60 mg daily, and ≤ 1/6 subjects experience a DLT at 40 mg daily, then 40 mg daily will be considered the RP2D. The dose of pembrolizumab will be constant at 200 mg IV every 3 weeks.
Time Frame: Throughout Cycle 1, up to 21 days
Population: There were 8 total patients enrolled in phase I cohorts of the study (5 in cohort 1 (PEM 200/CABO 40) and 3 in cohort 2 (PEM 200/CABO 60). Among the 5 patients in cohort 1, only 3 were evaluable for DLT and MTD. In total, 6 patients in phase I were evaluable for DLT and MTD.
Measure: Number; unit: mg
Groups:
- Phase 1: Pembrolizumab 200 mg IV Q3W Plus Cabozantinib 40mg or 60 mg PO QD: Pembrolizumab 200 mg intravenous (IV) infusion on day 1 of each 21-day cycle in combination with cabozantinib 40 mg or 60 mg orally once daily until disease progression, unacceptable toxicity, or consent withdrawal.
  Cabozantinib: Pharmaceutical form: tablets Route of administration: oral
  Pembrolizumab: Pharmaceutical form: solution Route of administration: injection
Arm/Group | Phase 1: Pembrolizumab 200 mg IV Q3W Plus Cabozantinib 40mg or 60 mg PO QD
Number analyzed (Participants) | 6
mg | 60

3. Secondary Outcome: Dose Limiting Toxicities
Description: Assessed through Common Terminology Criteria for Adverse Events (CTCAE) v 4.0. Dose Limiting Toxicity (DLT) was defined as any of the following events occurring during the DLT assessment window (21 days) and is assessed by the investigator to be likely related to study treatment (pembrolizumab and/or cabozantinib).
  * Grade ≥ 3 non-hematologic, non-hepatic adverse events
  * Grade 3 nausea, vomiting, or diarrhea lasting >72 hours despite maximal medical therapy.
  * Grade ≥ 4 neutropenia (ANC < 500 cells/μL) lasting > 7 days
  * Grade ≥ 3 febrile neutropenia
  * Grade ≥ 4 anemia
  * Grade ≥ 4 thrombocytopenia, or Grade 3 thrombocytopenia associated with clinically significant bleeding
  * Grade ≥ 3 elevation of serum hepatic transaminase (ALT or AST).
  * Grade ≥ 3 elevation of serum total bilirubin.
  * ALT or AST > 3 × upper limit of normal (ULN) AND total bilirubin >2 × ULN will require permanent treatment discontinuation.
Time Frame: Throughout Cycle 1, up to 21 days
Population: Total patients enrolled in phase I of the study who were evaluable for DLTs.
Measure: Number; unit: events
Groups:
- Phase 1 Cohort 1: Pembrolizumab 200 mg Plus Cabozantinib 40mg: Pembrolizumab 200 mg intravenous (IV) infusion on day 1 of each 21-day cycle in combination with cabozantinib 40 mg orally once daily until disease progression, unacceptable toxicity, or consent withdrawal.
  Cabozantinib: Pharmaceutical form: tablets Route of administration: oral
  Pembrolizumab: Pharmaceutical form: solution Route of administration: injection
- Phase 1 Cohort 2: Pembrolizumab 200 mg Plus Cabozantinib 60mg: Pembrolizumab 200 mg intravenous (IV) infusion on day 1 of each 21-day cycle in combination with cabozantinib 60 mg orally once daily until disease progression, unacceptable toxicity, or consent withdrawal.
  Cabozantinib: Pharmaceutical form: tablets Route of administration: oral
  Pembrolizumab: Pharmaceutical form: solution Route of administration: injection
Arm/Group | Phase 1 Cohort 1: Pembrolizumab 200 mg Plus Cabozantinib 40mg | Phase 1 Cohort 2: Pembrolizumab 200 mg Plus Cabozantinib 60mg
Number analyzed (Participants) | 3 | 3
events | 0 | 0

4. Secondary Outcome: Progression-Free Survival
Description: Measured as the time it takes for an occurrence of documented disease progression. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Beginning of study to end of study, or death, whichever comes first, up to 5 years
Population: All 40 patients treated at the RP2D were included in the survival analyses.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- All Patients Treated at the RP2D of Pembrolizumab 200 mg IM Q3W Plus Cabozantinib 60 mg PO QD: Pembrolizumab 200 mg intravenous (IV) infusion on day 1 of each 21-day cycle in combination with cabozantinib at the RP2D orally once daily for up to 35 cycles, until disease progression, unacceptable toxicity, or consent withdrawal. All participants who stop pembrolizumab after 35 cycles with SD or better may be eligible for up to an additional 17 cycles (approximately 1 year) of pembrolizumab treatment if they progress after stopping pembrolizumab from the initial treatment phase.
  Cabozantinib: Pharmaceutical form: tablets Route of administration: oral
  Pembrolizumab: Pharmaceutical form: solution Route of administration: injection
Arm/Group | All Patients Treated at the RP2D of Pembrolizumab 200 mg IM Q3W Plus Cabozantinib 60 mg PO QD
Number analyzed (Participants) | 40
months | 10.45 [6.25 to 14.63]

5. Secondary Outcome: Overall Survival
Description: Measured as the time it takes for an occurrence of death due to any cause
Time Frame: Beginning of study to end of study, or death, whichever comes first, up to 5 years
Population: All 40 patients treated at the RP2D were included in the survival analyses.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | All Patients Treated at the RP2D of Pembrolizumab 200 mg IM Q3W Plus Cabozantinib 60 mg PO QD
Number analyzed (Participants) | 40
months | 30.81 [24.23 to 40]

6. Secondary Outcome: Disease Control Rate (DCR), AKA Clinical Benefit Rate (CBR)
Description: DCR is the sum of the complete response, partial response, and stable disease rates
Time Frame: Beginning of study to end of study, or death, whichever comes first, up to 5 years
Population: All Evaluable Patients Treated at Pembrolizumab 200 mg IV Q3W + Cabozantinib 60 mg PO QD
Measure: Number (95% Confidence Interval); unit: % of patients
Groups:
- All Evaluable Patients Treated at Pembrolizumab 200 mg IV Q3W + Cabozantinib 60 mg PO QD: Pembrolizumab 200 mg intravenous (IV) infusion on day 1 of each 21-day cycle in combination with cabozantinib at the RP2D orally once daily for up to 35 cycles, until disease progression, unacceptable toxicity, or consent withdrawal. All participants who stop pembrolizumab after 35 cycles with SD or better may be eligible for up to an additional 17 cycles (approximately 1 year) of pembrolizumab treatment if they progress after stopping pembrolizumab from the initial treatment phase.
  Cabozantinib: Pharmaceutical form: tablets Route of administration: oral
  Pembrolizumab: Pharmaceutical form: solution Route of administration: injection
Arm/Group | All Evaluable Patients Treated at Pembrolizumab 200 mg IV Q3W + Cabozantinib 60 mg PO QD
Number analyzed (Participants) | 38
% of patients | 97.4 [86.5 to 99.9]

7. Secondary Outcome: Duration of Response
Description: Duration of time that patients maintain RECIST response to treatment
Time Frame: Time of first response as measured by RECIST 1.1 to time of progression or death, whichever comes first, up to 5 years
Population: All patients evaluable for response at the RP2D of Pembrolizumab 200 mg IM Q3W plus Cabozantinib 60 mg PO QD
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | All Patients Treated at the RP2D of Pembrolizumab 200 mg IM Q3W Plus Cabozantinib 60 mg PO QD
Number analyzed (Participants) | 38
months | 8.3 [4.6 to 15.1]

ADVERSE EVENTS:
Time Frame: 5 yrs and 3 months
Arm/Group | Phase 1: Pembrolizumab 200 mg Plus Cabozantinib 40mg | Phase 1: Pembrolizumab 200 mg Plus Cabozantinib 60mg | Phase 2: Pembrolizumab 200 mg Plus Cabozantinib at the RP2D
All-Cause Mortality (participants affected / at risk) | 5/5 | 2/3 | 24/37
Serious Adverse Events (participants affected / at risk) | 2/5 | 2/3 | 17/37
Other Adverse Events (participants affected / at risk) | 5/5 | 3/3 | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Pembrolizumab 200 mg Plus Cabozantinib 40mg (N=5) | Phase 1: Pembrolizumab 200 mg Plus Cabozantinib 60mg (N=3) | Phase 2: Pembrolizumab 200 mg Plus Cabozantinib at the RP2D (N=37)
GI bleed (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Increased cancer related pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Intestinal Pneumatosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Duodenal Hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Pembrolizumab 200 mg Plus Cabozantinib 40mg (N=5) | Phase 1: Pembrolizumab 200 mg Plus Cabozantinib 60mg (N=3) | Phase 2: Pembrolizumab 200 mg Plus Cabozantinib at the RP2D (N=37)
Abdominal Distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 4 (6)
Abdominal Pain (Gastrointestinal disorders) | 2 (5) | 0 (0) | 16 (22)
Alkaline Phosphatase increased (Investigations) | 1 (1) | 0 (0) | 7 (9)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 11 (22)
Anorexia (Metabolism and nutrition disorders) | 2 (3) | 2 (3) | 24 (30)
Anxiety (Psychiatric disorders) | 1 (2) | 0 (0) | 5 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 17 (22)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 12 (17)
Chills (General disorders) | 1 (1) | 0 (0) | 8 (9)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (3) | 16 (18)
Cough (Reproductive system and breast disorders) | 2 (4) | 1 (1) | 15 (20)
Creatinine increased (Investigations) | 2 (2) | 2 (3) | 6 (8)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 2 (5) | 25 (75)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 9 (11)
Dysgeusia (Nervous system disorders) | 2 (6) | 2 (2) | 20 (31)
Enlarged preauricular node (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 2 (2) | 1 (1) | 12 (16)
Fatigue (General disorders) | 4 (6) | 3 (4) | 17 (42)
Fever (General disorders) | 1 (5) | 0 (0) | 12 (13)
Dark Stool (Gastrointestinal disorders) | 1 (1) | 0 (0) | 5 (9)
Soft stool (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1 (3) | 1 (1) | 10 (16)
Diaphragm tightness (General disorders) | 1 (1) | 0 (0) | 1 (1)
Lightheaded (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (6) | 11 (17)
Bumps under tongue (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus irritation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (3) | 3 (3)
Generalized weakness (General disorders) | 1 (1) | 1 (1) | 9 (10)
Necrotic nasal septum (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 3 (4)
Hypertension (Cardiac disorders) | 1 (1) | 1 (1) | 16 (26)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 6 (12)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (4) | 2 (9) | 18 (50)
Gout (Infections and infestations) | 1 (3) | 0 (0) | 0 (0)
Increased INR (Investigations) | 1 (1) | 0 (0) | 0 (0)
Elevated C-Telopeptide Beta-Crossed-Linked Serum (Investigations) | 1 (1) | 0 (0) | 0 (0)
Irregular menstruation (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 1 (1) | 17 (32)
Bilateral Femoral pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
nail discoloration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 13 (19)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 24 (45)
Foot hyperesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 1 (1) | 6 (7)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (6) | 18 (37)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 1 (1) | 2 (3)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 4 (4)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2 (6) | 2 (2) | 13 (24)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 10 (16)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (2) | 15 (34)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 4 (4)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Nasal ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (4) | 0 (0)
Vaginal itching/burning (Reproductive system and breast disorders) | 1 (2) | 0 (0) | 2 (3)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 7 (8)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Urinary urgency/ (Renal and urinary disorders) | 2 (3) | 1 (1) | 4 (6)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (5)
Raynaud's (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Voice alteration (General disorders) | 1 (1) | 1 (1) | 11 (11)
Watering eyes (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Weight loss (Metabolism and nutrition disorders) | 3 (3) | 3 (4) | 25 (38)
Vomitting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 16 (35)
Aspartate aminotransferase increased (Hepatobiliary disorders) | 0 (0) | 2 (6) | 18 (26)
Adrenal insufficiency (Endocrine disorders) | 0 | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 3 (4) | 17 (32)
Allergic Reaction (Immune system disorders) | 0 (0) | 1 (1) | 1 (2)
Polycythemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0)
Elevated lactate dehydrogenase (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 1 (1) | 4 (4)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 9 (12)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 15 (20)
Dysphasia (Nervous system disorders) | 0 (0) | 1 (1) | 8 (9)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 14 (18)
Perichondritis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Edema face (General disorders) | 0 (0) | 1 (1) | 4 (4)
Diabetes mellitus Type II (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Flank pain (General disorders) | 0 (0) | 1 (1) | 2 (2)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 3 (5)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 9 (14)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (2) | 14 (21)
Strep Throat (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 1 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (4) | 6 (6)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Oral dysesthesia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 5 (5)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 14 (17)
Hair depigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 10 (10)
tinea corporis - umbilicus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Mouth Sensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 7 (7)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 6 (7)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) | 3 (3)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 6 (8)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 6 (6)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 2 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 10 (14)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 10 (12)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 8 (9)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 11 (13)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 10 (12)
hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (13)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 9 (15)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 5 (8)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 10 (11)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 9 (18)
Pain (general) (General disorders) | 0 (0) | 0 (0) | 22 (52)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 10 (17)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Tooth Infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (5)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 5 (6)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 2 (3)
Abnormal urinalysis (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Activity Change (General disorders) | 0 (0) | 0 (0) | 3 (5)
Blood Tinged Sputum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
body aches (General disorders) | 0 (0) | 0 (0) | 2 (2)
Callus on feet (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (4)
Chest pain (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Cold Intolerance (General disorders) | 0 (0) | 0 (0) | 5 (5)
colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Concentration Impairment (General disorders) | 0 (0) | 0 (0) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 6 (6)
Dental problems (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (6)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Diaphoresis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (5)
Duodenal Hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Elevated TSH (Endocrine disorders) | 0 (0) | 0 (0) | 3 (3)
Enterocolitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (4)
Finger Cramping (General disorders) | 0 (0) | 0 (0) | 3 (3)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (4)
Flu like symptoms (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Viral hepatitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Malaise (General disorders) | 0 (0) | 0 (0) | 3 (3)
Dysphoric Mood (Psychiatric disorders) | 0 (0) | 0 (0) | 4 (4)
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 3 (13)
Visual disturbances (Eye disorders) | 0 (0) | 0 (0) | 3 (3)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 5 (7)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (4)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Neck stiffness (General disorders) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-06-17): https://cdn.clinicaltrials.gov/large-docs/22/NCT03149822/Prot_SAP_ICF_000.pdf